CLINICAL TRIAL: NCT01651403
Title: A Randomized, Double-Blind Evaluation of the Antiviral Efficacy, Safety, and Tolerability of Tenofovir Disoproxil Fumarate Versus Placebo in Pediatric Patients With Chronic Hepatitis B Infection
Brief Title: Study to Evaluate the Antiviral Efficacy, Safety and Tolerability of Tenofovir Disoproxil Fumarate Versus Placebo in Pediatric Participants With Chronic Hepatitis B Infection
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-174-0144; 2012-000586-20 (EudraCT Number); 2024-517526-26 (Other: CTIS Number)
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tenofovir DF (Blinded Randomized Treatment) (Experimental): Participants will receive tenofovir disoproxil fumarate (tenofovir DF; TDF) for 72 weeks (protocol amendment 2) or 48 weeks (protocol amendment 3).
  Interventions: Drug: Tenofovir DF
- Placebo to match TDF (Blinded Randomized Treatment) (Placebo Comparator): Participants will receive TDF placebo for 72 weeks (protocol amendment 2) or 48 weeks (protocol amendment 3).
  Interventions: Drug: TDF Placebo
- Tenofovir DF (Open-label Treatment) (Experimental): Following 72 weeks (protocol amendment 2) or 48 weeks (protocol amendment 3) of blinded randomized treatment, participants will switch to open-label TDF treatment for an additional 120 weeks (protocol amendment 2) or 144 weeks (protocol amendment 3).
  Interventions: Drug: Tenofovir DF
- Tenofovir DF (Open-label Extension Phase) (Experimental): Following the completion of study at Week 192, participants may have the option to receive open-label TDF until it is commercially available in that country for treatment of chronic HBV in participants of their age and weight.
  Interventions: Drug: Tenofovir DF

INTERVENTIONS:
Drug: Tenofovir DF — * Participants weighing ≥ 17 kg will receive TDF one tablet administered orally once daily (150, 200, 250 or 300 mg tablets based on body weight).
  * Participants weighing < 17 kg or ≥ 17 kg who are unable to swallow a tablet will receive TDF oral powder in a dose of 8 mg/kg once daily up to a maximum dose of 300 mg.
  Other Names: Viread®
  Arms: Tenofovir DF (Blinded Randomized Treatment); Tenofovir DF (Open-label Extension Phase); Tenofovir DF (Open-label Treatment)
Drug: TDF Placebo — * Participants weighing ≥ 17 kg will receive TDF placebo tablet administered orally once daily.
  * Participants weighing < 17 kg or ≥ 17 kg who are unable to swallow a tablet will receive TDF placebo oral powder once daily.
  Arms: Placebo to match TDF (Blinded Randomized Treatment)

SUMMARY:
The primary objective of this study is to evaluate the antiviral efficacy of tenofovir disoproxil fumarate (tenofovir DF; TDF) versus placebo in pediatric population (aged 2 to < 12 years at the time of enrollment) with chronic hepatitis B (CHB) infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or Female, 2 to < 12 years of age
* Weight ≥ 10 kg
* Chronic HBV infection ≥ 6 months
* Hepatitis B e antigen (HBeAg)-positive or HBeAg-negative
* HBV Viral Load ≥ 100,000 copies/mL
* Alanine aminotransferase (ALT) ≥ 1.5 x the upper limit of the normal range (ULN) at screening
* Creatinine Clearance ≥ 80 mL/min/1.73m^2
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3, hemoglobin ≥ 10 g/dL
* Negative pregnancy test at screening
* No prior tenofovir DF therapy (participants may have received prior interferon-alfa and/or other oral anti-HBV nucleoside/nucleotide therapy; participants must have discontinued interferon-alfa therapy ≥ 6 months prior to screening; participants experienced on other anti-HBV nucleoside/nucleotide therapy must have discontinued therapy ≥ 16 weeks prior to screening to avoid flare if randomized to the placebo arm)

Key Exclusion Criteria:

* Pregnant or lactating
* Decompensated liver disease
* Received interferon therapy within 6 months of screening
* Received anti-HBV nucleoside/nucleotide therapy within 16 weeks of screening
* Alpha-fetoprotein levels > 50 ng/mL
* Evidence of hepatocellular carcinoma (HCC)
* Co-infection with human immunodeficiency virus (HIV), acute hepatitis A virus (HAV), hepatitis C virus (HCV), or hepatitis D virus (HDV)
* Chronic liver disease not due to HBV
* History of significant renal, cardiovascular, pulmonary, neurological or bone disease
* Long term non-steroidal, anti-inflammatory drug therapy

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2027-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (21):
- United States (5):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
- India (6):
  - Nirmal Hospital Private Limited, Surat, Gujarat
  - Medanta -The Medicity, Gurgaon, Haryana
  - Colors Children Hospital, Nagpur, Maharashtra
  - SMS Medical College and Hospital, Jaipur, Rajasthan
  - M.V. Hospital and Research Centre 314/30 Mirza Mandi Chowk, Lucknow, Uttar Pradesh
  - St. John Hospital & Medical Center, Bangalore
- Romania (3):
  - Grigore Alexandrescu Emergency Clinical Hospital for Children, Bucharest
  - Fundeni Clinical Institute - Constantinesco, Bucharest
  - Victor Babes Clinical Hospital of Infectious Diseases and Pneumophtisology, Craiova
- South Korea (5):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Kyungpook National University, Daegu
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Children's Hospital, Seoul
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Result] (Oral Presentation) Mei-Hwei Chang, Jae Hong Park, Jorge A. Bezerra, Daniela Pacura, Sandeep Nijhawan, Byung-Ho Choe, et al. Randomized, Double-Blind, Placebo-Controlled Trial of Tenofovir Disoproxil Fumarate (TDF) in Children with Chronic Hepatitis B (CHB). Hepatology, 2018; 68 (Suppl 1): 49A.
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-174-0144

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Asia, and Europe.The first participant was screened on 06 December 2012. The last Week 192 study visit occurred on 02 June 2020.
Pre-assignment Details: 176 participants were screened.
Groups:
- Tenofovir Disoproxil Fumarate: Blinded Randomized Phase: Tenofovir disoproxil fumarate (TDF) tablet or oral powder once daily (up to 300 mg depending on weight) for 72 weeks (protocol amendment 2) or 48 weeks (protocol amendment 3)
  Open-Label Treatment Phase: After Week 72 (protocol amendment 2) or Week 48 (protocol amendment 3), participants switched to open-label TDF treatment for an additional 120 weeks (protocol amendment 2) or 144 weeks (protocol amendment 3).
  Open-Label Extension Phase: After Week 192, participants are offered open-label TDF treatment until it was commercially available in that country for treatment of chronic HBV in individuals of their age and weight.
- Placebo: Blinded Randomized Phase: Placebo tablet or oral powder once daily for 72 weeks (protocol amendment 2) or 48 weeks (protocol amendment 3)
  Open-Label Treatment Phase: After Week 72 (protocol amendment 2) or Week 48 (protocol amendment 3), participants switched to open-label TDF treatment for an additional 120 weeks (protocol amendment 2) or 144 weeks (protocol amendment 3).
  Open-Label Extension Phase: After Week 192, participants are offered open-label TDF treatment until it was commercially available in that country for treatment of chronic HBV in individuals of their age and weight.
Period: Double-Blind Period (Through Week 48/72)
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo
Started | 60 | 30
Completed | 56 | 25
Not Completed | 4 | 5
Not completed — Participant Noncompliance | 1 | 1
Not completed — Withdrew Consent/Assent | 3 | 3
Not completed — Randomized but not Treated | 0 | 1
Period: Open-Label Phase (Weeks 49/73-192)
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo
Started | 56 | 25
Completed | 35 | 11
Not Completed | 21 | 14
Not completed — Continuing Study | 13 | 9
Not completed — Investigator decision | 2 | 1
Not completed — Withdrew consent/assent | 6 | 4

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all randomized participants who received at least 1 dose of study drug. Participants were analyzed according to the treatment they actually received during the double-blind phase.
Groups:
- Tenofovir Disoproxil Fumarate: Blinded Randomized Phase: TDF tablet or oral powder once daily (up to 300 mg depending on weight) for 72 weeks (protocol amendment 2) or 48 weeks (protocol amendment 3)
  Open-Label Treatment Phase: After Week 72 (protocol amendment 2) or Week 48 (protocol amendment 3), participants switched to open-label TDF treatment for an additional 120 weeks (protocol amendment 2) or 144 weeks (protocol amendment 3).
  Open-Label Extension Phase: After Week 192, participants are offered open-label TDF treatment until it was commercially available in that country for treatment of chronic HBV in individuals of their age and weight.
- Total: Total of all reporting groups
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo | Total
Number analyzed (Participants) | 60 | 29 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 6 (2.5) | 7 (3.2) | 6 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 12 | 39
  Male | 33 | 17 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 60 | 29 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 41 | 17 | 58
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 15 | 11 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 23 | 11 | 34
  Romania | 13 | 10 | 23
  United States | 14 | 3 | 17
  Taiwan | 2 | 0 | 2
  India | 8 | 5 | 13
HBV DNA [Mean (Standard Deviation); unit: log10 IU/mL] | 8.089 (0.7208) | 8.133 (1.2538) | 8.103 (0.9214)
Hepatitis B Virus Surface Antigen (HBsAg) [Count of Participants; unit: Participants]
  Positive | 60 | 29 | 89
  Negative | 0 | 0 | 0
Hepatitis B e antigen (HBeAg) [Count of Participants; unit: Participants]
  Positive | 56 | 29 | 85
  Negative | 4 | 0 | 4
HBeAb [Count of Participants; unit: Participants]
  Positive | 4 | 0 | 4
  Negative or Missing | 56 | 29 | 85
Spine Bone Mineral Density [Mean (Standard Deviation); unit: g/cm^2] | 0.586 (0.1196) | 0.626 (0.1567) | 0.599 (0.1332)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum HBV DNA < 400 Copies/mL (69 IU/mL) at Week 48 (Missing = Failure Approach)
Time Frame: Week 48
Population: The Full Analysis Set (FAS) included randomized participants who have received at least 1 dose of study drug. Participants will be analyzed according to the treatment to which they were randomized. The missing equals failure approach was used where all participants with missing data were considered to have failed to achieve the endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- TDF (Blinded Randomized Phase): Blinded Randomized Phase: TDF tablet or oral powder once daily (up to 300 mg depending on weight) for 72 weeks (protocol amendment 2) or 48 weeks (protocol amendment 3)
- Placebo (Blinded Randomized Phase): Blinded Randomized Phase: Placebo tablet or oral powder once daily for 72 weeks (protocol amendment 2) or 48 weeks (protocol amendment 3)
Arm/Group | TDF (Blinded Randomized Phase) | Placebo (Blinded Randomized Phase)
Number analyzed (Participants) | 60 | 29
percentage of participants | 76.7 [64.0 to 86.6] | 6.9 [0.8 to 22.8]
Statistical Analysis 1: Comparison: TDF (Blinded Randomized Phase) vs Placebo (Blinded Randomized Phase); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; 2-sided Cochran-Mantel-Haenszel test adjusted for age at baseline and region strata
Statistical Analysis 2: Comparison: TDF (Blinded Randomized Phase) vs Placebo (Blinded Randomized Phase); Test type: Superiority; p < 0.001, Fisher Exact; Fisher's exact test without adjusting for strata at baseline

2. Secondary Outcome: Percentage of Participants With Hepatitis B e Antigen (HBeAg) Seroconversion at Week 48
Description: HBeAg seroconversion was defined as HBeAg loss and a change from HBeAb negative or missing at baseline to HBeAb positive.
Time Frame: Week 48
Population: Serologically Evaluable FAS For HBeAg loss/seroconversion: participants who were randomized and had received at least 1 dose of study drug, and with HBeAg positive and HBeAb negative or missing at baseline. The missing equals failure approach was used where all participants with missing data were considered to have failed to reach the endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | TDF (Blinded Randomized Phase) | Placebo (Blinded Randomized Phase)
Number analyzed (Participants) | 56 | 29
percentage of participants | 25.0 | 24.1
Statistical Analysis 1: Comparison: TDF (Blinded Randomized Phase) vs Placebo (Blinded Randomized Phase); Test type: Superiority; p = 0.935, Cochran-Mantel-Haenszel; 2-sided Cochran-Mantel-Haenszel test adjusted for age at baseline and region strata

3. Secondary Outcome: Percentage of Participants With Normal Alanine Aminotransferase (ALT) at Week 48, Based on the American Association for the Study of Liver Diseases (AASLD) Normal Range
Description: Normal ALT was defined as ≤ 30 U/L for males and females 0-12 years based on the AASLD pediatric normal range.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed. The missing equals failure approach was used where all participants with missing data were considered to have failed to reach the endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | TDF (Blinded Randomized Phase) | Placebo (Blinded Randomized Phase)
Number analyzed (Participants) | 60 | 29
percentage of participants | 51.7 | 17.2
Statistical Analysis 1: Comparison: TDF (Blinded Randomized Phase) vs Placebo (Blinded Randomized Phase); Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; 2-sided Cochran-Mantel-Haenszel tests adjusted for age at baseline and region strata

4. Secondary Outcome: Percentage of Participants With Normal ALT at Week 192, Based on the AASLD Normal Range
Description: Normal ALT was defined as ≤ 30 U/L for males and females 0-12 years based on the AASLD pediatric normal range.
Time Frame: Week 192
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- TDF to TDF: Blinded Randomized Phase: TDF tablet or oral powder once daily (up to 300 mg depending on weight) for 72 weeks (protocol amendment 2) or 48 weeks (protocol amendment 3)
  Open-Label Treatment Phase: After Week 72 (protocol amendment 2) or Week 48 (protocol amendment 3), participants switched to open-label TDF treatment for an additional 120 weeks (protocol amendment 2) or 144 weeks (protocol amendment 3).
- Placebo to TDF: Blinded Randomized Phase: Placebo tablet or oral powder once daily for 72 weeks (protocol amendment 2) or 48 weeks (protocol amendment 3)
  Open-Label Treatment Phase: After Week 72 (protocol amendment 2) or Week 48 (protocol amendment 3), participants switched to open-label TDF treatment for an additional 120 weeks (protocol amendment 2) or 144 weeks (protocol amendment 3).
Arm/Group | TDF to TDF | Placebo to TDF
Number analyzed (Participants) | 60 | 29
percentage of participants | 71.7 | 51.7

5. Secondary Outcome: Percentage of Participants With Normal ALT at Week 48, Based on the Central Lab Normal Range
Description: Normal ALT was defined as ≤ 34 U/L for females aged 2-15 years old or males aged 1-9 years old, and ≤ 43 U/L for males aged 10-15 years old based on the central lab normal range.
Time Frame: Week 48
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | TDF (Blinded Randomized Phase) | Placebo (Blinded Randomized Phase)
Number analyzed (Participants) | 60 | 29
percentage of participants | 65.0 | 17.2
Statistical Analysis 1: Comparison: TDF (Blinded Randomized Phase) vs Placebo (Blinded Randomized Phase); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; 2-sided Cochran-Mantel-Haenszel tests adjusted for age at baseline and region strata

6. Secondary Outcome: Percentage of Participants With Normal ALT at Week 192, Based on the Central Lab Normal Range
Description: as for outcome 5
Time Frame: Week 192
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | TDF to TDF | Placebo to TDF
Number analyzed (Participants) | 60 | 29
percentage of participants | 80.0 | 62.1

7. Secondary Outcome: Percentage of Participants With Normalized ALT at Week 48, Based on the AASLD Normal Range
Description: Normal ALT was defined as ≤ 30 U/L for males and females 0-12 years based on the AASLD pediatric normal range. ALT normalization was defined as an ALT value that changed from above the normal range at baseline to within the normal range at the given postbaseline visit.
Time Frame: Week 48
Population: Participants in the Full Analysis Set with abnormal ALT values at baseline were analyzed. The missing equals failure approach was used where all participants with missing data were considered to have failed to reach the endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | TDF (Blinded Randomized Phase) | Placebo (Blinded Randomized Phase)
Number analyzed (Participants) | 60 | 28
percentage of participants | 51.7 | 17.9
Statistical Analysis 1: Comparison: TDF (Blinded Randomized Phase) vs Placebo (Blinded Randomized Phase); Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; 2-sided Cochran-Mantel-Haenszel tests adjusted for age at baseline and region strata

8. Secondary Outcome: Percentage of Participants With Normalized ALT at Week 192, Based on the AASLD Normal Range
Description: as for outcome 7
Time Frame: Week 192
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | TDF to TDF | Placebo to TDF
Number analyzed (Participants) | 60 | 28
percentage of participants | 71.7 | 50.0

9. Secondary Outcome: Percentage of Participants With Normalized ALT at Week 48, Based on the Central Lab Normal Range
Description: Normal ALT was defined as ≤ 34 U/L for females aged 2-15 years old or males aged 1-9 years old, and ≤ 43 U/L for males aged 10-15 years old based on the central lab normal range. ALT normalization was defined as an ALT value that changed from above the normal range at baseline to within the normal range at the given postbaseline visit.
Time Frame: Week 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | TDF (Blinded Randomized Phase) | Placebo (Blinded Randomized Phase)
Number analyzed (Participants) | 58 | 27
percentage of participants | 65.5 | 14.8
Statistical Analysis 1: Comparison: TDF (Blinded Randomized Phase) vs Placebo (Blinded Randomized Phase); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; 2-sided Cochran-Mantel-Haenszel tests adjusted for age at baseline and region strata

10. Secondary Outcome: Percentage of Participants With Normalized ALT at Week 192, Based on the Central Lab Normal Range
Description: as for outcome 9
Time Frame: Week 192
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | TDF to TDF | Placebo to TDF
Number analyzed (Participants) | 58 | 27
percentage of participants | 79.3 | 59.3

11. Secondary Outcome: Composite Endpoint of Percentage of Participants With HBV DNA < 400 Copies/mL (69 IU/mL) and Normalized ALT (Based on AASLD Normal Range) at Week 48
Description: as for outcome 7
Time Frame: Week 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | TDF (Blinded Randomized Phase) | Placebo (Blinded Randomized Phase)
Number analyzed (Participants) | 60 | 28
percentage of participants | 46.7 | 7.1
Statistical Analysis 1: Comparison: TDF (Blinded Randomized Phase) vs Placebo (Blinded Randomized Phase); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; 2-sided Cochran-Mantel-Haenszel tests adjusted for age at baseline and region strata

12. Secondary Outcome: Composite Endpoint of Percentage of Participants With HBV DNA < 400 Copies/mL (69 IU/mL) and Normalized ALT (Based on AASLD Normal Range) at Week 192
Description: as for outcome 7
Time Frame: Week 192
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | TDF to TDF | Placebo to TDF
Number analyzed (Participants) | 60 | 28
percentage of participants | 70.0 | 42.9

13. Secondary Outcome: Composite Endpoint of Percentage of Participants With HBV DNA < 400 Copies/mL (69 IU/mL) and Normalized ALT (Based on Central Lab Normal Range) at Week 48
Description: as for outcome 9
Time Frame: Week 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | TDF (Blinded Randomized Phase) | Placebo (Blinded Randomized Phase)
Number analyzed (Participants) | 58 | 27
percentage of participants | 53.4 | 7.4
Statistical Analysis 1: Comparison: TDF (Blinded Randomized Phase) vs Placebo (Blinded Randomized Phase); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; 2-sided Cochran-Mantel-Haenszel tests adjusted for age at baseline and region strata

14. Secondary Outcome: Composite Endpoint of Percentage of Participants With HBV DNA < 400 Copies/mL (69 IU/mL) and Normalized ALT (Based on Central Lab Normal Range) at Week 192
Description: as for outcome 9
Time Frame: Week 192
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | TDF to TDF | Placebo to TDF
Number analyzed (Participants) | 58 | 27
percentage of participants | 75.9 | 55.6

15. Secondary Outcome: Percentage of Participants With HBV DNA < 169 Copies/mL (29 IU/mL) at Week 48
Time Frame: Week 48
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | TDF (Blinded Randomized Phase) | Placebo (Blinded Randomized Phase)
Number analyzed (Participants) | 60 | 29
percentage of participants | 71.7 | 6.9
Statistical Analysis 1: Comparison: TDF (Blinded Randomized Phase) vs Placebo (Blinded Randomized Phase); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; two-sided Cochran-Mantel-Haenszel test adjusted for age at baseline and region strata

16. Secondary Outcome: Percentage of Participants With HBV DNA < 169 Copies/mL (29 IU/mL) at Week 192
Time Frame: Week 192
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | TDF to TDF | Placebo to TDF
Number analyzed (Participants) | 60 | 29
percentage of participants | 81.7 | 62.1

17. Secondary Outcome: Percentage of Participants With HBsAg Loss at Week 48
Description: HBsAg Loss was defined as a change from HBsAg positive or missing at baseline to HBsAg negative.
Time Frame: Week 48
Population: Serologically Evaluable Full Analysis Set For HBsAg Loss/Seroconversion; The missing equals failure approach was used where all participants with missing data were considered to have failed to reach the endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | TDF (Blinded Randomized Phase) | Placebo (Blinded Randomized Phase)
Number analyzed (Participants) | 60 | 29
percentage of participants | 3.3 | 3.4
Statistical Analysis 1: Comparison: TDF (Blinded Randomized Phase) vs Placebo (Blinded Randomized Phase); Test type: Superiority; p > 0.999, Cochran-Mantel-Haenszel; Two-sided Cochran-Mantel-Haenszel test adjusted for age at baseline and region strata

18. Secondary Outcome: Percentage of Participants With HBsAg Loss at Week 192
Description: HBsAg Loss was defined as a change from HBsAg positive or missing at baseline to HBsAg negative.
Time Frame: Week 192
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | TDF to TDF | Placebo to TDF
Number analyzed (Participants) | 60 | 29
percentage of participants | 10.0 | 0

19. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion at Week 48
Description: HBsAg seroconversion was defined as HBsAg loss and a change from HBsAb negative or missing at baseline to HBsAb positive.
Time Frame: Week 48
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | TDF (Blinded Randomized Phase) | Placebo (Blinded Randomized Phase)
Number analyzed (Participants) | 60 | 29
percentage of participants | 0 | 0

20. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion at Week 192
Description: as for outcome 19
Time Frame: Week 192
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | TDF to TDF | Placebo to TDF
Number analyzed (Participants) | 60 | 29
percentage of participants | 0 | 0

21. Secondary Outcome: Number of Participants With Sequence Changes From Baseline Within the HBV Polymerase for Participants Who Were Viremic (HBV DNA ≥ 400 Copies/mL [69 IU/mL]) Including Participants With Confirmed Virologic Breakthrough at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with serum samples available at baseline and with HBV DNA ≥ 69 IU/mL at Week 48 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | TDF (Blinded Randomized Phase) | Placebo (Blinded Randomized Phase)
Number analyzed (Participants) | 10 | 26
Participants | 5 | 7

22. Secondary Outcome: Number of Participants With Sequence Changes From Baseline Within the HBV Polymerase for Participants Who Were Viremic (HBV DNA ≥ 400 Copies/mL [69 IU/mL]) Including Participants With Confirmed Virologic Breakthrough at Week 96
Time Frame: Baseline; Week 96
Population: Participants in the Full Analysis Set with serum samples available at baseline and with HBV DNA ≥ 69 IU/mL at Week 96 were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- TDF to TDF: Blinded Randomized Phase: Tenofovir disoproxil fumarate (TDF) tablet or oral powder once daily (up to 300 mg depending on weight) for 72 weeks (protocol amendment 2) or 48 weeks (protocol amendment 3)
  Open-Label Treatment Phase: After Week 72 (protocol amendment 2) or Week 48 (protocol amendment 3), participants switched to open-label TDF treatment for an additional 120 weeks (protocol amendment 2) or 144 weeks (protocol amendment 3).
Arm/Group | TDF to TDF | Placebo to TDF
Number analyzed (Participants) | 5 | 12
Participants | 1 | 2

23. Secondary Outcome: Number of Participants With Sequence Changes From Baseline Within the HBV Polymerase for Participants Who Were Viremic (HBV DNA ≥ 400 Copies/mL [69 IU/mL]) Including Participants With Confirmed Virologic Breakthrough at Week 144
Time Frame: Baseline; Week 144
Population: Participants in the Full Analysis Set with serum samples available at baseline and with HBV DNA ≥ 69 IU/mL at Week 144 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | TDF to TDF | Placebo to TDF
Number analyzed (Participants) | 4 | 1
Participants | 1 | 0

24. Secondary Outcome: Number of Participants With Sequence Changes From Baseline Within the HBV Polymerase for Participants Who Were Viremic (HBV DNA ≥ 400 Copies/mL [69 IU/mL]) Including Participants With Confirmed Virologic Breakthrough at Week 192
Time Frame: Baseline; Week 192
Population: Participants in the Full Analysis Set with serum samples available at baseline and with HBV DNA ≥ 69 IU/mL at Week 192 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | TDF to TDF | Placebo to TDF
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

25. Secondary Outcome: Percentage of Participants With ≥ 4% Decrease From Baseline in Spine Bone Mineral Density (BMD) at Week 48
Time Frame: Baseline; Week 48
Population: Spine Dual X-Ray Absorptiometry (DXA) Analysis Set: all randomized participants who received at least 1 dose of study drug and had nonmissing baseline spine bone mineral density values.
Measure: Number; unit: percentage of participants
Arm/Group | TDF (Blinded Randomized Phase) | Placebo (Blinded Randomized Phase)
Number analyzed (Participants) | 60 | 29
percentage of participants | 18.3 | 6.9
Statistical Analysis 1: Comparison: TDF (Blinded Randomized Phase) vs Placebo (Blinded Randomized Phase); Test type: Other — Comparison of the difference in percentages; Exact Chan-Zhang method = 11.4, 95% CI 2-sided [-6.9 to 25.1]

26. Secondary Outcome: Percentage of Participants With ≥ 4% Decrease From Baseline in Spine BMD at Week 192
Time Frame: Baseline; Week 192
Population: Participants in the Spine DXA Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF to TDF | Placebo to TDF
Number analyzed (Participants) | 60 | 29
percentage of participants | 18.3 | 6.9
Statistical Analysis 1: Comparison: TDF to TDF vs Placebo to TDF; Test type: Other — Comparison of the difference in percentages; Exact Chan-Zhang method = 11.4, 95% CI 2-sided [-6.9 to 25.1]

27. Secondary Outcome: Percent Change From Baseline in BMD of Spine at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Spine DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change in spine BMD
Arm/Group | TDF (Blinded Randomized Phase) | Placebo (Blinded Randomized Phase)
Number analyzed (Participants) | 55 | 25
Percent change in spine BMD | 3.798 (5.9118) | 7.557 (4.9790)
Statistical Analysis 1: Comparison: TDF (Blinded Randomized Phase) vs Placebo (Blinded Randomized Phase); Test type: Superiority; p = 0.007, ANOVA; two-sided superiority test

28. Secondary Outcome: Percent Change From Baseline in BMD of Spine at Week 192
Time Frame: Baseline; Week 192
Population: Participants in the Spine DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change in spine BMD
Arm/Group | TDF to TDF | Placebo to TDF
Number analyzed (Participants) | 52 | 18
Percent change in spine BMD | 19.168 (12.2805) | 26.085 (14.2586)

29. Primary Outcome: Percentage of Participants With Serum HBV DNA < 400 Copies/mL (69 IU/mL) at Week 48 (Missing = Excluded Approach)
Time Frame: Week 48
Population: Participants in the Full Analysis Set with available data were analyzed. The missing equals failure approach was used where all participants with missing data were excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TDF (Blinded Randomized Phase) | Placebo (Blinded Randomized Phase)
Number analyzed (Participants) | 55 | 26
percentage of participants | 83.6 [71.2 to 92.2] | 7.7 [0.9 to 25.1]
Statistical Analysis 1: Comparison: TDF (Blinded Randomized Phase) vs Placebo (Blinded Randomized Phase); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; 2-sided Cochran-Mantel-Haenszel test adjusted for age at baseline and region strata

ADVERSE EVENTS:
Time Frame: First dose date up to the Week 192 Data Cut for Open-Label Phase; Additional adverse event data will be reported after study is completed and final analysis is done.
Description: Safety Analysis all randomized participants who have received at least 1 dose of study drug. Participants were analyzed according to the treatment to which they received during the blinded phase. All-cause mortality: The Randomized Analysis Set included all participants who were randomized into the study.
Groups:
- TDF to TDF (Open-Label Phase); Placebo to TDF (Open-Label Phase): Open-Label Treatment Phase: After Week 72 (protocol amendment 2) or Week 48 (protocol amendment 3), participants switched to open-label TDF treatment for an additional 120 weeks (protocol amendment 2) or 144 weeks (protocol amendment 3).
  Open-Label Extension Phase: After Week 192, participants are offered open-label TDF treatment until it was commercially available in that country for treatment of chronic HBV in individuals of their age and weight.
Arm/Group | TDF (Blinded Randomized Phase) | Placebo (Blinded Randomized Phase) | TDF to TDF (Open-Label Phase) | Placebo to TDF (Open-Label Phase)
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/30 | 0/56 | 0/25
Serious Adverse Events (participants affected / at risk) | 10/60 | 2/29 | 8/56 | 3/25
Other Adverse Events (participants affected / at risk) | 38/60 | 16/29 | 21/56 | 7/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TDF (Blinded Randomized Phase) (N=60) | Placebo (Blinded Randomized Phase) (N=29) | TDF to TDF (Open-Label Phase) (N=56) | Placebo to TDF (Open-Label Phase) (N=25)
Acute hepatitis B (Infections and infestations) | 1 | 0 | 0 | 0
Adenovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TDF (Blinded Randomized Phase) (N=60) | Placebo (Blinded Randomized Phase) (N=29) | TDF to TDF (Open-Label Phase) (N=56) | Placebo to TDF (Open-Label Phase) (N=25)
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 0 | 2
Pyrexia (General disorders) | 9 | 2 | 4 | 0
Ear infection (Infections and infestations) | 3 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 9 | 2 | 12 | 1
Otitis media (Infections and infestations) | 3 | 1 | 1 | 1
Pharyngitis (Infections and infestations) | 3 | 3 | 2 | 1
Tonsillitis (Infections and infestations) | 3 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 9 | 5 | 3 | 3
Varicella (Infections and infestations) | 3 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 3 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (7):
  • Study Protocol: Original (2011-07-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT01651403/Prot_000.pdf
  • Study Protocol: Amendment 1 (2012-03-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT01651403/Prot_001.pdf
  • Study Protocol: Amendment 2 (2012-11-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT01651403/Prot_002.pdf
  • Study Protocol: Amendment 3 (2016-02-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT01651403/Prot_003.pdf
  • Study Protocol: Amendment 4 (2016-08-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT01651403/Prot_004.pdf
  • Statistical Analysis Plan: Week 48 Analysis (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT01651403/SAP_005.pdf
  • Statistical Analysis Plan: Week 192 Analysis (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT01651403/SAP_006.pdf